CLINICAL TRIAL: NCT04323111
Title: Evaluation of Metzenbaum Technique in Correction of Caudal End Nasal Septal Deviation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Madonna Atef Aziz, resident at ENT department at assiut university hospital, Assiut University
Other Study IDs: metzenbaum in caudal end NSD
Record Dates: First submitted 2020-03-22; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Nasal Septal Caudal Dislocation
Keywords: caudal end nasal septal deviation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: metzenbaum's technique — surgical procedure for correction of caudal end nasal septal deviation

SUMMARY:
• To evaluate the results of Metzenbaum 's technique in correction of the Caudal end septal deviation on nasal airway obstruction

DETAILED DESCRIPTION:
Deviation of Nasal septum in different parts may have various functional or aesthetic effects . The etiology of a deviated septum is generally congenital, but may also be as a result of trauma or iatrogenic causes. Most important is the Caudal septal deviation which narrows the airway and impairs major mechanisms supporting the tip, leading to tip-ptosis and airway collapse. .The correction of caudal septal deviations can be a challenging problem so many techniques have been described and tested to correct caudal septal deflections . Attempts to correct nasal septal deformities were described in the medical literature as early as the late 19th century , and till now there is not one specific technique that is agreed upon by surgeons worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Assiut University Clinic of Otolaryngology department.
* Aging from 16 to 45 years old
* Patients complaining of nasal airway obstruction causes by caudal septal deviation.

Exclusion Criteria:

* Other causes of airway obstruction e.g. nasal polyps, hypertrophied inferior turbinates'
* External nasal deformities
* Contraindications for general anesthesia

Ages: 16 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: all adults having nasal airway obstruction due to caudal end nasal septal deviation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
the caudal end deviation of the nasal septum corrected is measured by photographic documentation | 6 month
  Photographs will be taken in the 6 dimensional (frontal,basal, lateral and oblique) views of the nose at two points ,First photograph set will be taken in preoperative period. The second photograph set will taken at six months follow up. Both these photographs will be shown to the patient and he/she was asked to give a score to rate the difference in appearance on a 4 point scale 4 point scale for evaluating postoperative outcome
  1. Little/no photographic evidence of residual caudal septal deviation.
  2. Marked improvement but was still detectable by careful observation.
  3. Mild improvement/not improved.
  4. Made worse after surgical intervention.
air way obstruction which will be be evaluated by The Nasal Obstruction Symptom Evaluation (NOSE) scale score questionnaire | 2 month
  The Nasal Obstruction Symptom Evaluation (NOSE) scale score is a questionnaire that each patient will take to compare the symptoms of air way obstruction improvement after surgery . the patients will take it at two points , first in pre - operative assessment and second in post operative follow up after 2 month

REFERENCES:
- [Background] Chandra RK, Patadia MO, Raviv J. Diagnosis of nasal airway obstruction. Otolaryngol Clin North Am. 2009 Apr;42(2):207-25, vii. doi: 10.1016/j.otc.2009.01.004. PMID 19328887
- [Background] Lal D, Corey JP. Acoustic rhinometry and its uses in rhinology and diagnosis of nasal obstruction. Facial Plast Surg Clin North Am. 2004 Nov;12(4):397-405, v. doi: 10.1016/j.fsc.2004.04.002. PMID 15337107
- [Background] Menegat F, Monnazzi MS, Silva BN, de Moraes M, Gabrielli MA, Pereira-Filho VA. Assessment of nasal obstruction symptoms using the NOSE scale after surgically assisted rapid maxillary expansion. Int J Oral Maxillofac Surg. 2015 Nov;44(11):1346-50. doi: 10.1016/j.ijom.2015.06.018. Epub 2015 Jul 15. PMID 26187045
- [Background] Haack J, Papel ID. Caudal septal deviation. Otolaryngol Clin North Am. 2009 Jun;42(3):427-36. doi: 10.1016/j.otc.2009.03.005. PMID 19486740
- [Background] Sedwick JD, Lopez AB, Gajewski BJ, Simons RL. Caudal septoplasty for treatment of septal deviation: aesthetic and functional correction of the nasal base. Arch Facial Plast Surg. 2005 May-Jun;7(3):158-62. doi: 10.1001/archfaci.7.3.158. PMID 15897403
- [Background] Batioglu-Karaaltin A, Yigit O, Donmez Z. A new persistent suture technique for correction of caudal septal dislocation. J Craniofac Surg. 2014 Nov;25(6):2169-71. doi: 10.1097/SCS.0000000000000893. PMID 25329853